CLINICAL TRIAL: NCT04797364
Title: Pharmacogenetic Supported Prescribing in Kids
Acronym: PGx-SParK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Chad Bousman, Associate Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: REB20-0900
Record Dates: First submitted 2021-03-09; First posted 2021-03-15 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Mental Health Impairment
Keywords: Child; Adolescent; Mental Health; Psychiatry; Pharmacogenetics; Depression; Anxiety; OCD; Psychosis; Bipolar Disorder
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders; Psychotic Disorders; Bipolar Disorder | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacogenetic Testing (Experimental): Pharmacogenetic testing panel (CYP2B6, CYP2C9, CYP2C19, CYP2D6, CYP3A5, NUDT15, SLCO1B1, TPMT, VKORC1)
  Interventions: Diagnostic Test: Pharmacogenetic Testing

INTERVENTIONS:
Diagnostic Test: Pharmacogenetic Testing — Participants will donate a 2ml (teaspoon) sample of saliva. DNA extracted from the saliva sample will be used for genotyping. Genotyping results will be translated into an interpretative clinical report using evidence-based software (Sequence2Script) developed by our group and delivered to the treating physician for use in their clinical decision-making. The report will contain genotyping results, predicted phenotype, and evidence-based drug selection and dosing recommendations relevant to the child's current and future care

SUMMARY:
Implementation of pharmacogenetic testing for children and adolescents aged 6-24 who are starting or changing psychiatric medication.

DETAILED DESCRIPTION:
Children with moderate to severe mental health conditions (e.g. depression, anxiety, OCD) or neurodevelopmental disorders (e.g., autism spectrum disorders, ADHD) are frequently prescribed medications as either the sole form of treatment or in combination with psychotherapy. However, up to 50% of these children will not respond or experience burdensome adverse drug reactions to these medications. Current use of mental health-related medications (e.g., antidepressants, antipsychotics) in children can be best described as a trial-and-error process that can impact the well-being of those taking the medications and their families at a considerable economic cost. However, this trial-and-error process could, in part, be avoided through the application of pharmacogenetic testing, a specific type of genetic testing that has the potential to improve drug efficacy and reduce the morbidity, mortality and cost associated with adverse drug reactions. The aim of this project is to implement and evaluate an evidence-based pharmacogenetic testing service to improve drug treatment outcomes in children receiving mental health care.

Our objectives are to:

1. Implement Canada's first pharmacogenetics testing service to improve drug treatment outcomes in children receiving mental health care.
2. Collect performance, outcome, and economic indicators related to the pharmacogenetics testing service.
3. Establish a research platform for the discovery of new genetic and non-genetic markers of drug treatment outcomes relevant to mental health care in children.

ELIGIBILITY:
Inclusion Criteria:

* Medical records available
* The initiation, change, dose adjustment, or augmentation of psychiatric medication(s) is indicated
* Treating psychiatrist, family physician, or pediatrician licensed in Alberta, British Columbia, Saskatchewan, or Manitoba requests pharmacogenetic testing

Exclusion Criteria:

* Medically unstable or lacking capacity to provided informed consent
* Unwillingness of child to provide saliva sample for genetic analysis
* History of liver or bone marrow (hematopoietic cell) transplant

Ages: 6 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6000 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Adverse drug reactions | 6-months
  Relative change in adverse drug reaction frequency
Symptom severity | 6-months
  Relative change in symptom severity

SECONDARY OUTCOMES:
Healthcare utilization | 6-months
  Relative change in healthcare utilization

CONTACTS AND LOCATIONS:
Overall Officials: Chad Bousman, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Bharthi K, Zuberi R, Maruf AA, Shaheen SM, McCloud R, Heintz M, McAusland L, Arnold PD, Bousman CA. Impact of Cytochrome P450 Genetic Variation on Patient-Reported Symptom Improvement and Side Effects Among Children and Adolescents Treated with Fluoxetine. J Child Adolesc Psychopharmacol. 2024 Feb;34(1):21-27. doi: 10.1089/cap.2023.0039. PMID 38377520